CLINICAL TRIAL: NCT05998148
Title: Patient Reported Outcomes From Patients Seen in Virtual Phone Visits Compared to In-Person Physical Visits for Post-Operative Follow-Up at a Sports Medicine Clinic: A Prospective Randomized Controlled Trial
Brief Title: Virtual Phone Visits Compared to In-Person Physical Visits for Post-Operative Follow-Up at a Sports Medicine Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonathan Wu (Other)
Responsible Party: Sponsor-Investigator, Jonathan Wu, Researcher, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Organization: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 18CR-32251-01
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Results first posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Patient Satisfaction; Sports Injury; Surgery; Orthopedic Disorder
Keywords: patient reported outcomes; telemedicine; virtual; phone; sports medicine; in person
MeSH Terms: conditions — Patient Satisfaction; Athletic Injuries; Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard in-person appointment visits (No Intervention): Randomly selected participants will receive standard in-person post-operative appointment visits at 6 week, 12 week, and 6 months after surgery.
- virtual phone appointment visits (Experimental): Randomly selected participants will receive virtual telemedicine post-operative appointment visits at 6 week, 12 week, and 6 months after surgery.
  Interventions: Other: virtual phone appointment visits

INTERVENTIONS:
Other: virtual phone appointment visits — Patient will have post-operative appointments that place with telemedicine. The visits will will be virtual phone appointments scheduled at approximately 6 weeks, 12 weeks, and 6 months after surgery.
  Arms: virtual phone appointment visits

SUMMARY:
This study will compare patient reported outcomes (PROs) of patients seen at virtual phone visits compared to in-person visits for 6 weeks, 12 weeks, and 6 months post-operative follow up at a sports medicine clinic. This study will determine if there is a difference in PROs between these two groups of patients. The investigators hypothesize patients who are seen during a virtual phone visit will report different PRO compared to patients who are seen during an in-person visit for post-operative follow-up at 6-months.

DETAILED DESCRIPTION:
In this prospective study, the investigators will enroll patients undergoing operative intervention at a Sports Medicine clinic.

The patient will arrive at a pre-operative clinic appointment, surgery, or 2 week post-operative appointment to sign the consent form in the presence of study team member and a witness in order to be eligible to participate in the study.

After consent is obtained, the Participant will be randomized to either in-person follow up or virtual phone follow up to take place after the 2-week post-op visit.

The randomization process will utilize block randomization and be conducted by an online program called http://www.randomization.com. The Participant will be assigned a number based on the order the Participant is enrolled in the study and that number will be randomly assigned to a follow-up group based on that number.

The Participant will be notified at the 2-week post-op or after if they will receive will in-person follow up or virtual phone follow-up. If the Participant in the virtual phone group feel they need an in-person visit, the Participant will be free to make an in-person follow-up. After each follow up visit (6-week, 12-week, and 6-month), the Participant will be asked to fill out 30-minute surveys.

The surveys the Participant will be asked to fill out are the following:

1. Knee Injury and Osteoarthritis Outcome Score (KOOS JR)- a knee specific survey
2. Oxford Shoulder Outcome Measure
3. Patient Reported Outcomes Measurement Information system (PROMIS) Global
4. General Health Questionnaires (2)
5. Patient Satisfaction Survey -The investigators will have the patient complete this also after every visit to see if their preferences change over time as their recovery changes.

If a Participant attends an in-person post-operative follow up visit, then the study team member will check to see if the participant is on the in-person list. If the participant is on the list, then he or she will be given a tablet to fill out the online survey after the appointment. The tablet will be set up so a link to the surveys can be accessed and participants can fill out the surveys. The surveys are on REDCaps (https://research.lundquist.org/redcap/surveys/?s=NK3YH4NWL3). Participants will be able to fill out the survey at home because the survey will be emailed to the participant. For Participants that attend a virtual appointment, an online link to the survey on REDCap will be sent to the Participant's email. Members of the study team can also call participant from both arms to conduct the survey over the phone.

The first page of the survey asks for the Participant's name, date of birth, and preferred language (English or Spanish), how comfortable filling out the form, who is completing the form, which joints, amount of pain, and amount of back pain. The next page of the survey will be a joint specific survey and will depend on the joint selected on the first page and the language chosen. It can be the KOOS JR, Oxford Shoulder Outcome Measure, or PROMIS Global. There is a separate patient satisfaction survey that the patient will complete.

Participants will have appointments at the sports clinic for suture removal (10 to 14 days after surgery), and evaluation at 6 weeks, 12 weeks, and 6 months after surgery per usual practice.

Study coordinator will check the upcoming Participant schedule and ensure the correct appointment is scheduled.

The source records that will be used to collect data about the Participants are the surveys, type of surgery, and results of follow-up visits. The data collected will be asked on the surveys which include demographic information- Participants' injury region, age, gender, and time since operative intervention.

A participant registry will be maintained on an excel spreadsheet to maintain participant's contact information, appointment schedule, and completion of surveys. The registry will also track which participant is in the in-person arm or virtual arm. After a new participant is consented, the information is added to the participant registry. Participant appointment dates will be kept on the registry. Each appointment scheduled in the electronic medical record will be entered in the registry and track the progress of the participant. If there is a patient that requires a change in intervention group, that is marked on the registry. For participants that do not follow up or are lost to follow up, that information is recorded.

For missing data, the information will be kept for data analysis for intention to treat analysis. The participants with missing data will be removed to conduct per protocol analysis.

Statistical analysis will be conducted to compare the total scores of each survey results from participants in the in-person group with participants in the virtual phone group. Each Participant's outcome scores will be averaged and standard deviation calculated.

Participant outcomes scores from the 6 month visit will be compared across the in-patient group and virtual phone group using Student t-test. Statistical significance will be based on an α level of 0.05.

The PROMIS Global-Physical is used to calculate the required sample size as it as the largest range of the outcome measures resulting in the most conservative estimates.

For a statistical significance of 0.05, Power of 80%, and assuming a large effect size of 0.61, 34 Participants are required per group for a total of 68 Participants.

The investigators will attempt to recruit at least 104 Participants. This will allow room in case of patients are removed or fall from the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants are at least 18 years of age.
* Participants who are seen at Harbor-UCLA Medical Center sports medicine clinic.
* Participants have agreed to have operative intervention.
* Participants must own a phone with reliable calling capabilities.
* The Participants must have access to reliable internet to fill out the online survey.
* The Participants must be able to provide consent.
* Participants may include pregnant patients.

Exclusion Criteria:

* Patients that are under the age of 18
* any cognitive impaired adult
* any adult unable to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P Andrawis, M.D., Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Locations (1):
- Harbor-UCLA Medical Center, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data that results in a publication will be made available upon request.
Time Frame: information will be made available starting after publication. The information will be available for 3 years after publication.
Access Criteria: Criteria include other researchers interested in patient reported outcomes, for analyses related to telemedicine. Study coordinator will review requests for more data.

REFERENCES:
- [Background] Sharareh B, Schwarzkopf R. Effectiveness of telemedical applications in postoperative follow-up after total joint arthroplasty. J Arthroplasty. 2014 May;29(5):918-922.e1. doi: 10.1016/j.arth.2013.09.019. Epub 2013 Dec 15. PMID 24342278
- [Background] Grandizio LC, Foster BK, Klena JC. Telemedicine in Hand and Upper-Extremity Surgery. J Hand Surg Am. 2020 Mar;45(3):239-242. doi: 10.1016/j.jhsa.2019.09.007. Epub 2019 Nov 9. PMID 31718846
- [Background] Preston N, McHugh GA, Hensor EMA, Grainger AJ, O'Connor PJ, Conaghan PG, Stone MH, Kingsbury SR. Developing a standardized approach to virtual clinic follow-up of hip and knee arthroplasty. Bone Joint J. 2019 Aug;101-B(8):951-959. doi: 10.1302/0301-620X.101B8.BJJ-2018-1566.R1. PMID 31362551

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started in March 2022 and ended in March 2023. The location of recruitment was a sports medicine clinic at a county hospital.
Pre-assignment Details: There are no significant events that occur after participant enrollment, but prior to assignment of participants to an arm or group.
Groups:
- Virtual Phone Appointment Visits: Randomly selected patients will receive virtual telemedicine post-operative appointment visits at 6 week, 12 week, and 6 months after surgery.
- Standard In-person Appointment Visits: Randomly selected participants will attend standard in-person post-operative appointment visits at 6 week, 12 week, and 6 months after surgery.
Period: Allocation
Arm/Group | Virtual Phone Appointment Visits | Standard In-person Appointment Visits
Started | 48 | 42
Completed | 47 | 38
Not Completed | 1 | 4
Not completed — Did not attend any appointments | 1 | 4
Period: Follow-Up
Arm/Group | Virtual Phone Appointment Visits | Standard In-person Appointment Visits
Started | 47 | 38
Completed | 45 | 35
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Change in insurance | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Standard In-person Appointment Visits: Randomly selected patients will receive standard in-person post-operative appointment visits at 6 week, 12 week, and 6 months after surgery.
- Total: Total of all reporting groups
Arm/Group | Virtual Phone Appointment Visits | Standard In-person Appointment Visits | Total
Number analyzed (Participants) | 45 | 35 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] — The age is determined by the age of the patient at the time of enrollment.
  years | 43.6 (15.98) | 41.83 (13.26) | 42.82 (14.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 31 | 21 | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Racial identity is self-selected by the patient
  Participants
    Racial Identity: Hispanic | 24 | 26 | 50
    Racial Identity: Caucasian | 12 | 3 | 15
    Racial Identity: Black | 5 | 4 | 9
    Racial Identity: Asian | 4 | 2 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45 | 35 | 80
Primary Language [Count of Participants; unit: Participants] — Primary language is self selected by the patient
  Participants
    English | 39 | 17 | 56
    Spanish | 6 | 18 | 24
Type of Surgery [Count of Participants; unit: Participants]
  Knee | 27 | 26 | 53
  Shoulder | 18 | 9 | 27

OUTCOME MEASURES:

1. Primary Outcome: PROMIS Physical and Mental Scores
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) GLOBAL Survey is divided into PROMIS Physical and PROMIS Mental. Minimum score 16.2, Maximum Score 67.2 for PROMIS Physical. Minimum score 21.2, Maximum score 67.6 for PROMIS Mental. Higher score means better outcome.
Time Frame: 6 month post-operative visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Phone Appointment Visits | Standard In-person Appointment Visits
Number analyzed (Participants) | 45 | 35
score on a scale
  PROMIS Physical | 50.46 (7.84) | 50.26 (7.76)
  PROMIS Mental | 56.51 (10.02) | 60.21 (8.47)
Statistical Analysis 1: Comparison: Virtual Phone Appointment Visits vs Standard In-person Appointment Visits; The null hypothesis states that the virtual group and in-person group exhibit no difference in mean PROMIS physical score. From the literature, an effect size of 0.618 was obtained from the PROMIS physical. Using a power of 80% and a significance level of 0.05, it was determined that a sample size of 34 per group would detect a statistical difference between the groups. An intention-to-treat analysis was conducted on the scores at the 6-month follow-up appointment; Test type: Other; p = 0.91, t-test, 2 sided — The threshold for statistical significance was p= 0.05; Since 2 hypothesis tests are conducted, we applied a Bonferroni correction. Our new adjusted threshold level is 0.05/2= 0.025; Mean Difference (Net) = 0.2 — Treatment Difference = Virtual - Standard In-person
Statistical Analysis 2: Comparison: Virtual Phone Appointment Visits vs Standard In-person Appointment Visits; The null hypothesis states that the virtual group and in-person group exhibit no difference in mean PROMIS mental score. The minimum sample size determined for the PROMIS physical score was applied to this outcome score. An intention-to-treat analysis was conducted on the scores at the 6-month follow-up appointment; Test type: Other; p = 0.077, t-test, 2 sided — The threshold for statistical significance was p= 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -3.7 — Treatment Difference = Virtual - Standard In-person
Statistical Analysis 3: Comparison: Virtual Phone Appointment Visits vs Standard In-person Appointment Visits; The null hypothesis states that the virtual group and in-person group exhibit no difference in mean PROMIS physical score. From the literature, effect size of 0.618 was obtained from PROMIS physical. Using a power of 80% and a significance level of 0.05, it was determined that a sample size of 34 per group would detect a statistical difference between the groups. A per-protocol analysis was conducted on the scores at the 6-month follow-up appointment. There were 34 patients in each group; Test type: Other; p = 0.75, t-test, 2 sided; Mean Difference (Net) = 0.56 — Treatment Difference = Virtual - Standard In-person
Statistical Analysis 4: Comparison: Virtual Phone Appointment Visits vs Standard In-person Appointment Visits; The null hypothesis states that the virtual group and in-person group exhibit no difference in mean PROMIS mental score. The minimum sample size determined for the PROMIS physical score was used for this analysis. A per-protocol analysis was conducted on the scores at the 6-month follow-up appointment. There were 34 patients in each group; Test type: Other; p = 0.049, t-test, 2 sided — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -4.49 — Treatment Difference = Virtual - Standard In-person

2. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score for Joint Replacement
Description: Survey scores from Knee injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS JR) for knee injuries. Minimum score 0. Max score 100. Higher score is better.
Time Frame: 6 month post-operative visit
Population: Only patients who underwent operative management on their knees filled out this survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Phone Appointment Visits | Standard In-person Appointment Visits
Number analyzed (Participants) | 27 | 26
score on a scale | 72.25 (17.69) | 68.41 (22.85)
Statistical Analysis 1: Comparison: Virtual Phone Appointment Visits vs Standard In-person Appointment Visits; There were 27 patients in the virtual phone group. There were 26 patients in the standard in-person group; Test type: Other; p = 0.49, t-test, 2 sided — The threshold for statistical significance was p=0.05; Mean Difference (Net) = 3.84 — Treatment Difference = Virtual - Standard In-person

3. Secondary Outcome: Oxford Shoulder Score
Description: Survey scores from the Oxford Shoulder score for shoulder injuries. Minimum is 0. Maximum is 48. Higher score is better.
Time Frame: 6 month post-operative visit
Population: Only participants who underwent operative management of their shoulder filled out this survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Phone Appointment Visits | Standard In-person Appointment Visits
Number analyzed (Participants) | 18 | 9
score on a scale | 35.65 (9.08) | 32 (15.33)
Statistical Analysis 1: Comparison: Virtual Phone Appointment Visits vs Standard In-person Appointment Visits; There are 18 patients in the virtual group. There are 9 patients in the standard in-person group; Test type: Other; p = 0.54, t-test, 2 sided — The threshold for statistical significance was p = 0.05; Mean Difference (Net) = 3.65 — Treatment Difference = Virtual - Standard In-person

4. Secondary Outcome: Patient Satisfaction Scores
Description: Patient satisfaction scores after in-person visit or virtual phone visit. Minium score is 1. Maximum Score 5. Higher score is better.
Time Frame: 6 month post-operative visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Phone Appointment Visits | Standard In-person Appointment Visits
Number analyzed (Participants) | 45 | 35
score on a scale | 4.5 (0.73) | 4.37 (0.60)
Statistical Analysis 1: Comparison: Virtual Phone Appointment Visits vs Standard In-person Appointment Visits; There are 45 patients in the virtual phone group. There are 35 patients in the standard in-person group; Test type: Other; p = 0.39, t-test, 2 sided — The threshold for statistical significance was p=0.05; Mean Difference (Net) = 0.13 — Treatment Difference = Virtual - Standard In-person

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Virtual Phone Appointment Visits | Standard In-person Appointment Visits
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/42
Other Adverse Events (participants affected / at risk) | 0/48 | 0/42

LIMITATIONS AND CAVEATS:
One of the limitations was the sample size. A second limitation was that we stopped recruitment at 90 patients because of time constraints instead of reaching the goal of 104 patients. A third limitation was the different methods which the virtual telemedicine visits took place. A fourth limitation was the different methods used to complete the surveys.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/48/NCT05998148/Prot_SAP_000.pdf